CLINICAL TRIAL: NCT03532217
Title: A Pilot Trial of Neoantigen DNA Vaccine in Combination With Nivolumab/Ipilimumab and PROSTVAC in Metastatic Hormone-Sensitive Prostate Cancer
Brief Title: Neoantigen DNA Vaccine in Combination With Nivolumab/Ipilimumab and PROSTVAC in Metastatic Hormone-Sensitive Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry); Prostate Cancer Foundation (Other); The Foundation for Barnes-Jewish Hospital (Other); Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201808043; CA209-9MW (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2018-04-25; First posted 2018-05-22 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer
MeSH Terms: interventions — PROSTVAC; Nivolumab; Ipilimumab; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PROSTVAC/Ipilimumab/Nivolumab/Neoantigen DNA vaccine (Experimental): * Within 60 days after the last chemo, patients will start a priming dose of PROSTVAC-V, and subsequent doses of PROSTVAC- F (weeks 0, 2, 5, 8, 11, 14, and 17). During "Treatment A" phase, subjects should receive nivolumab intravenously on Day 1 of each cycle every 3 weeks for 6 doses. Ipilimumab on Day 1 of each cycle every 3 weeks for 2 doses.
  * Patients will then receive a neoantigen DNA vaccine with continuous nivolumab treatment. The vaccine will be administered starting approximately week 21 by intramuscular injection for a total of 6 treatments every 28 days +/-7 days. Each DNA vaccination will be 4 mg vaccine administered intramuscularly using a TriGrid electroporation device. Patients will receive nivolumab at 480 mg every 28 days concurrently with neoantigen DNA vaccine. This is Treatment B. In the event the DNA vaccine production is delayed, patients will receive single agent nivolumab every 4 weeks beginning week 21 until the vaccine is ready
  Interventions: Biological: PROSTVAC-V; Biological: PROSTVAC-F; Drug: Nivolumab; Drug: Ipilimumab; Biological: Neoantigen DNA vaccine; Device: TriGrid Delivery System; Procedure: Tumor biopsy; Procedure: Peripheral blood; Procedure: Fecal samples; Procedure: Leukapheresis

INTERVENTIONS:
Biological: PROSTVAC-V — -Replication-competent vaccinia virus which has been engineered to encode the sequences for a modified human prostate-specific antigen (PSA) and a triad of co-stimulatory molecules (TRICOM)
Biological: PROSTVAC-F — -Fowlpox virus which does not replicate in human cells and has been engineered to encode the same sequences present in PROSTVAC-V.
Drug: Nivolumab — -Nivolumab is a human monoclonal antibody (mAb)
Drug: Ipilimumab — -Ipilimumab is a mAb blocking the inhibitory signal mediated by cytotoxic T Lymphocyte-associated antigen 4 (CTLA-4), a protein receptor that downregulates the immune system.
Biological: Neoantigen DNA vaccine — Each DNA vaccination will be 1 mL vaccine administered intramuscularly. At each vaccination time point, patients will receive two injections at separate sites.
Device: TriGrid Delivery System — -Electroporation device
  Other Names: TDS-IM
Procedure: Tumor biopsy — -Pre-treatment, post-treatment A (optional), and end of treatment
Procedure: Peripheral blood — -At the time of pre-treatment biopsy, mid-treatment of chemo-ADT, at time of enrollment (prior to POSTVAC administration), mid-treatment A, mid-treatment B (multiple)
Procedure: Fecal samples — -Post chemo/pre-treatment A, post-treatment A, pre-treatment B, post-treatment B
Procedure: Leukapheresis — * Post-treatment A/pre-treatment B
  * Mid-Treatment B, after Cycle 9 Day 1 and prior to Cycle 10 Day 1
  * End of treatment

SUMMARY:
This study study aims to elucidate the immune responses to a shared antigen vaccine (PROSTVAC) and tumor specific antigens generated DNA vaccine in combination with checkpoint blockade using nivolumab (anti-PD-1), and ipilimumab (anti-CTLA-4). Additionally, the investigators will study the impact of the combination immunotherapy on peripheral T cell activation, as well as immune response in the tumor microenvironment. Finally, the investigators will evaluate the safety and tolerability to this novel personalized immunotherapy in combination with checkpoint blockade.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* High risk/volume metastatic disease, as defined by 4 or more sites of disease or the presence of visceral metastases.
* Must have completed an adequate course of chemo-hormonal, first line therapy for metastatic hormone-sensitive prostate cancer, as determined by the investigator. Patients must remain on stable dose of ADT with castrate levels of testosterone (defined as testosterone < 50 ng/dL)
* At least 18 years of age.
* PSA may be undetectable after initial chemo-ADT.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 2,000/ul
  * Absolute neutrophil count ≥ 1,500/ul
  * Platelets ≥ 100,000/ul
  * Hemoglobin ≥ 9.0 g/ul
  * Total bilirubin ≤ 1.5 x ULN (except subjects with Gilbert's syndrome who must have a total bilirubin level of ≤ 3.0 ULN)
  * AST(SGOT) ≤ 3.0 x ULN
  * ALT(SGPT) ≤ 3.0 x ULN
  * Creatinine ≤ 1.5 x ULN OR calculated creatinine clearance ≥ 40 mL/min using the Cockcroft-Gault formula
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Must have a biopsy of a metastatic site of disease (may be archival) available and adequate for evaluation and determination of neoantigens by genomic analyses.
* Must have all AEs resolved to baseline prior to chemo-ADT, or if treatment related, resolved to grade 1 prior to enrollment.

Exclusion Criteria:

* Significant small cell or neuroendocrine component or histology, as determined by the institution's reading pathologist.
* Progression of disease as defined by a rising PSA (3 sequential values, at least 1 week apart) or radiographic progression based on RECIST1.1 or PCWG3 criteria.
* Prior treatment with a checkpoint inhibitor, neoantigen vaccine, or PROSTVAC.
* Participants with active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll.
* Diagnosis of atopic dermatitis or other active exfoliative skin condition
* History of concurrent second cancers requiring active, ongoing systemic treatment
* Currently receiving any other investigational agents.
* Known brain metastases. Prostate cancer patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis, and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to anti-PD-1, anti-CTLA-4, Prostvac-VF Tricom, DNA vaccines, or other agents used in the study.
* Prior allergy or significant systemic reaction to vaccinia.
* Prior reactions to monoclonal antibodies.
* Received hematopoietic stem cell transplant < 24 months prior to enrollment to this study, or received hematopoietic stem cell transplant ≥ 24 months prior to enrollment to this study but has graft-versus-host disease or disease relapse.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, clinically significant congestive heart failure (NYHA Class III, IV), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that in the opinion of the investigator would limit compliance with study requirements.
* Immunosuppressed status (e.g. HIV/AIDS, active HCV/HBV, high dose systemic steroids, etc.) as determined by the investigator; topical or inhaled steroids are acceptable.
* History of syncopal or vasovagal episode as determined by medical record and history in the 12 month period prior to first vaccination administration.
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for eligible injection sites (left and right medial deltoid region) exceeds 40 mm.
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art.
* Therapeutic or traumatic metal implant in the skin or muscle of either deltoid region.
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child.
* Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of regimen as defined by incidence of adverse events | Through 100 days after completion of treatment (estimated to be 55 weeks)
  -Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0
Immune response as measured by tetramers | Through completion of treatment (estimated to be 41 weeks)
  -MHC tetramers made against the identified neoantigens will be used to evaluate PBMC for neoantigen-reactive T cells
Immune response as measured by genomic studies | Through completion of treatment (estimated to be 41 weeks)
  -Laser capture microdissection will be performed to perform genomic studies on specific areas of tissue
Immune response as measured by flow cytometry | Through completion of treatment (estimated to be 41 weeks)
  -Multiparametric flow cytometry or CyTOF will be performed in parallel to evaluate for any shifts (in quality and quantity) in peripheral leukocyte subsets.
Safety and tolerability of regimen as defined by incidence of dose-limiting toxicities (DLTs) | Through 100 days after completion of treatment (estimated to be 55 weeks)
  -DLT is defined as any unexpected, treatment-related grade 4 or 5 adverse event that occurs with increased severity or incidence outside of known, expected toxicities, that occur in the first 6 patients enrolled (safety lead-in cohort)

SECONDARY OUTCOMES:
Failure-free survival (FFS) | Through completion of follow-up (estimated to be 65 weeks)
  -Defined as time from day 0 of treatment to evidence of at least one of the following: biochemical failure; radiographic or clinical progression either locally, in lymph nodes, or in distant metastases; or death from prostate cancer) compared to historical controls (ADT + docetaxel). Biochemical failure is defined as three consecutive rises (at lease one week apart) in PSA levels with the date of failure being the midpoint between the PSA nadir and the first PSA rise. Radiographic progression is defined as either RECIST1.1 or PCWG3 criteria.
Milestone survival | Through completion of follow-up (estimated to be 65 weeks)
  -Defined as the Kaplan-Meier survival probability
Number of participants who have PSA responses at 30% reduction level | Through completion of treatment (estimated to be 41 weeks)
  * Baseline PSA prior to start of treatment will be compared to PSA nadir during treatment and then the investigators can calculate how many participants hit 30% reduction from pretreatment levels
  * Participants who enroll with no detectable PSA will be considered not evaluable for this outcome measure
Number of participants who have PSA responses at 50% reduction level | Through completion of treatment (estimated to be 41 weeks)
  * Baseline PSA prior to start of treatment will be compared to PSA nadir during treatment and then the investigators can calculate how many participants hit 50% reduction from pretreatment levels
  * Participants who enroll with no detectable PSA will be considered not evaluable for this outcome measure
Radiographic progression as determined by RECIST 1.1 | Through completion of treatment (estimated to be 41 weeks)
  At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Radiographic progression as determined by Prostate Cancer Working Group 3 (PCWG3) | Through completion of treatment (estimated to be 41 weeks)
  * PCWG3 recommends that lymph nodes that were previously normal in size (< 1.0 cm) or pathologic in size must have grown by at least 5 mm in the short axis from baseline or nadir and be ≥ 1.0 cm in the short axis to be considered to have progressed. If the node progresses to ≥ 1.5 cm in the short axis, it is pathologic and measurable. Nodes that have progressed to between 1.0 and less than 1.5 cm are pathologic subject to clinical discretion and are nonmeasurable
  * The date of first metastasis is the date on which an unequivocal visceral lesion by RECIST 1.1 is determined
  * Documentation of radiographic evidence of metastatic disease should include the time of the unequivocal development of new sites on bone scintigraphy
Radiographic progression free survival (rPFS) | Through completion of treatment (estimated to be 41 weeks)
  -Radiographic progression-free survival (rPFS) is the time interval from baseline to the date when the first site of disease is found to progress (using a manifestation-specific definition of progression), or death, whichever occurs first. To better understand the effect of therapy on an individual site of disease, PCWG3 advises the date of progression in all specific sites be reported independently whether it is bone, nodes (pelvic or extrapelvic), visceral (lung, liver, adrenal, or CNS), or other.
Comparison of the immune correlates on matched tumor tissue and peripheral blood | Pre- and post-treatment (estimated to be 41 weeks)
  Laser capture microdissection will be performed to perform genomic studies on specific areas of tissue (eg tumor core, high TIL areas, tumor-stromal interface, etc). These will be correlated with multiplexed immunofluorescence studies, as well as assays on peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Pachynski, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu